CLINICAL TRIAL: NCT05363566
Title: Clinical Performance of the Baska MaskⓇ, the I-GelⓇ and the Self-Pressurized Air-QⓇ i
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-49-2021
Record Dates: First submitted 2022-03-19; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: The Baska Mask

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I (Active Comparator): will be inserted Single use supraglottic airway ( Baska mask® (proact Medical Ltd, Northants, UK)
  Interventions: Device: airway divice
- group II (Active Comparator): will be inserted Single use supraglottic airway ( I-gel® ) (Intersurgical Ltd, Wokingham, Berkshire, UK)
  Interventions: Device: airway divice
- group III (SP Air-Q) (n = 26) (Active Comparator): will be inserted Single use supraglottic airway (self-pressurized Air-Q intubating laryngeal airway (Air-Q SP®)) (Mercury Medical, Clearwater, FL, USA)
  Interventions: Device: airway divice

INTERVENTIONS:
Device: airway divice — inserted airway device

SUMMARY:
The Baska mask (proact Medical Ltd, Northants, UK) is the latest addition to an era of supraglottic airway devices in clinical use. It is made of medical grade silicone; it has many advantages in its constructions over other LMA, a cuff less membranous bowl in which the saliva secretion collected. An inbuilt "tab" that allows to extend its angulation for straightforward negotiation of the oropharyngeal curve during placement

ELIGIBILITY:
* Inclusion criteria

  1. Adult patients from 18 to 60 years of age.
  2. American Society of Anesthesiologists (ASA) physical status I and II
  3. Both genders
  4. Patients scheduled for elective surgeries lasting less than 2 hours under general anesthesia on spontaneous ventilation.
  5. El Ganzouri index Score ≥ 4
  6. Patients with BMI < 35 kg/m2
* Exclusion criteria

  1. The patients who will be refusal or inability to give informed consent,
  2. ASA class III or IV
  3. El Ganzouri index Score < 4,
  4. Oropharyngeal pathology making a proper SAD fit unlikely as weak dentation, neck pathology
  5. Respiratory illness including upper respiratory infection or pneumonia within the six weeks preceding surgery
  6. Risk for gastric aspiration (e.g., hiatus hernia, gastro-oesophageal reflux disease or non-fasting status), expected duration of surgery longer than 2 h
  7. Contraindication to SGA use including morbid obesity (body mass index 35 kg m-1, history of obstructive sleep apnea)
  8. Any condition for which the primary anesthesia team deemed intubation with a tracheal tube to be necessary.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-11-13 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
insertion time | 1 hour
  To determine the time taken for insertion of the device. (It will be calculated from the time of the mask will be taken away from the patient's face till the moment of the appearance of square wave capnography upstroke with the presence of sufficient ventilation) (second )

SECONDARY OUTCOMES:
Ease of device insertion | 1 hours
  will be graded using a five-point scoring system (4 = insertion at first attempt without tactile resistance, 3 = insertion at first attempt with little tactile resistance, 2 = insertion at first attempt with significant tactile resistance, 1 = insertion successful at second/third attempt, 0 = insertion failed at three attempts).
Oropharyngeal leak pressures | 1 hours
  Oropharyngeal leak pressures (OLPs) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working